CLINICAL TRIAL: NCT00489099
Title: A Study in Healthy Young Adults To Assess the Safety, Tolerability, and Immunogenicity of a Recombinant Hepatitis B Vaccine Manufactured by a Process Upgrade
Brief Title: A Research Study to Test Safety, Tolerability, and Immunogenicity of a Recombinant Hepatitis B Vaccine Manufactured With an Upgrade to the Production Process (V232-054)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: V232-054; 2007_565
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis B Infection
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- V232 Modified Process Hepatitis B Vaccine: Lot A (Experimental): Recombivax HB™ (Hepatitis B Vaccine [Recombinant]) modified process Lot A administered as a 1 mL intramuscular injection on Day 1, Month 1, and Month 6.
  Interventions: Biological: V232 Modified Process Hepatitis B Vaccine: Lot A
- V232 Modified Process Hepatitis B Vaccine: Lot B (Experimental): Recombivax HB™ (Hepatitis B Vaccine [Recombinant]) modified process Lot B administered as a 1 mL intramuscular injection on Day 1, Month 1, and Month 6.
  Interventions: Biological: V232 Modified Process Hepatitis B Vaccine: Lot B
- V232 Modified Process Hepatitis B Vaccine: Lot C (Experimental): Recombivax HB™ (Hepatitis B Vaccine [Recombinant]) modified process Lot C administered as a 1 mL intramuscular injection on Day 1, Month 1, and Month 6.
  Interventions: Biological: V232 Modified Process Hepatitis B Vaccine: Lot C
- V232 Current Process Hepatitis B Vaccine (Active Comparator): Recombivax HB™ (Hepatitis B Vaccine [Recombinant]) current process administered as a 1 mL intramuscular injection on Day 1, Month 1, and Month 6.
  Interventions: Biological: V232 Current Process Hepatitis B Vaccine

INTERVENTIONS:
Biological: V232 Modified Process Hepatitis B Vaccine: Lot A
  Arms: V232 Modified Process Hepatitis B Vaccine: Lot A
Biological: V232 Modified Process Hepatitis B Vaccine: Lot B
  Arms: V232 Modified Process Hepatitis B Vaccine: Lot B
Biological: V232 Modified Process Hepatitis B Vaccine: Lot C
  Arms: V232 Modified Process Hepatitis B Vaccine: Lot C
Biological: V232 Current Process Hepatitis B Vaccine
  Arms: V232 Current Process Hepatitis B Vaccine

SUMMARY:
A study to evaluate the safety, tolerability, and immunogenicity of a recombinant hepatitis B vaccine manufactured using an upgrade to the production process. The primary hypotheses tested at 1 month after the third dose of vaccine are the following: 1) the 3 lots of the process upgrade vaccine induce similar seroprotection rates to hepatitis B surface antigen (HBsAg), 2) the combined lots of the process upgrade vaccine induce adequate seroprotection to HBsAg, and 3) the process upgrade vaccine will induce geometric mean antibody titers to HBsAg that are non-inferior or superior to those induced by the current process vaccine.

ELIGIBILITY:
Inclusion Criteria:

* In general good health
* Female participants have a negative pregnancy test just prior to vaccination on Day 1

Exclusion Criteria:

* History of Hepatitis B Infection or vaccination
* Known or suspected hypersensitivity to any component of Recombivax HB™ vaccine (e.g., aluminum, yeast)
* Administration of hepatitis B immune globulin, serum immune globulin, or any other blood-derived product within 3 months prior to vaccination on Day 1
* Receipt of an inactivated virus vaccine within 14 days or a live virus vaccine within 30 days prior to vaccination on Day 1
* Participation on prior study using an investigational drug or vaccine in prior 3 months
* Known or suspected impairment of immunologic function or recent use of immunomodulatory medications, excluding topical or inhaled steroids
* Pregnant or nursing women or women planning to become pregnant within the study period

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 860 (Actual)
Dates: Start 2005-06; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Seroprotection to Hepatitis B Surface Antigen | 1 month after the third vaccination (Month 7)
Geometric Mean Titers to Hepatitis B Surface Antigen | 1 month after the third vaccination (Month 7)

SECONDARY OUTCOMES:
Percentage of Participants with an Adverse Experience | Up to 15 days after any vaccination
Percentage of Participants with an Injection-site Adverse Experience | Up to 15 days after any vaccination
Percentage of Participants with a Systemic Adverse Experience | Up to 15 days after any vaccination
Percentage of Participants with Fever (>=37.8°C, 100.0°F) | Up to 5 days after any vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Van Damme P, Minervini G, Liss CL, McCarson B, Vesikari T, Boslego JW, Bhuyan PK. Safety, tolerability and immunogenicity of a recombinant hepatitis B vaccine manufactured by a modified process in healthy young adults. Hum Vaccin. 2009 Feb;5(2):92-7. doi: 10.4161/hv.5.2.6587. Epub 2009 Feb 14. PMID 18690015
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html